CLINICAL TRIAL: NCT05476900
Title: A Randomized, Open-label, Multicenter, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HR19042 Capsules in the Treatment of Autoimmune Hepatitis.
Brief Title: A Study to Evaluate the Efficacy and Safety of HR19042 Capsules in the Treatment of Autoimmune Hepatitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR19042-202
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, multicenter, parallel groups, Phase II clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12 mg HR19042 Capsules QD (Experimental)
  Interventions: Drug: HR19042 Capsules
- 4 mg HR19042 Capsules TID (Experimental)
  Interventions: Drug: HR19042 Capsules
- 8 mg HR19042 Capsules QD (Experimental)
  Interventions: Drug: HR19042 Capsules

INTERVENTIONS:
Drug: HR19042 Capsules — HR19042 Capsules

SUMMARY:
This study will evaluate the efficacy and safety of HR19042 capsules for the treatment of autoimmune hepatitis. It will also explore the optimal frequency and dosage of HR19042 capsules administration for the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤Female or male patients≤70 years old；
2. Clinical-confirmed autoimmune hepatitis；
3. Biopsy-confirmed autoimmune hepatitis；
4. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥ 3 × upper limit of normal (ULN)；
5. Willing and able to give informed consent and follow the protocols during the trial.

Exclusion Criteria:

1. Patients with other chronic liver diseases；
2. Patients with liver cirrhosis；
3. Patients with hepatic encephalopathy；
4. Positive results in HIV-Ab/TP-Ab/hepatitis virus tests
5. Severe chronic or active infection requiring systemic anti-infective therapy within 14 days before screening；
6. Patients with severe cardiovascular diseases；
7. Patients with malignancy within the past 5 years；
8. Patients received organ transplantation；
9. Patients treated with any systemic corticosteroids within 3 months before screening；
10. Patients treated with any systemic immunosuppressive drugs within the 6 months before screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Percentage of biochemical response after 12 weeks of treatment. | 12 weeks

SECONDARY OUTCOMES:
Percentage of biochemical response with the absence of glucocorticoid-related adverse events after 12 weeks of treatment. | 12 weeks
Percentage of partial response after 12 weeks of treatment | 12 weeks
Percentage of biochemical response after 24 weeks of treatment. | 24 weeks
Percentage of biochemical response with the absence of glucocorticoid-related adverse events after 24 weeks of treatment. | 24 weeks
Percentage of partial response after 24 weeks of treatment. | 24 weeks
Change from baseline in serum ALT levels. | 2, 4, 8, 12, 18, 24 weeks
Change from baseline in serum AST levels. | 2, 4, 8, 12, 18, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided